CLINICAL TRIAL: NCT02706054
Title: Treatment of Recent Onset Low Back Pain With Periradicular Injections of Meloxicam: a Randomized, Double Blind, Placebo Controlled Cross-over Study
Brief Title: Treatment of Recent Onset Low Back Pain With Periradicular Injections of Meloxicam
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MELO-RCT
Record Dates: First submitted 2016-02-03; First posted 2016-03-11 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2016-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Sodium Chloride; Meloxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- C-group (Placebo Comparator): patients receiving an IM saline injection near the nerve root (periradicular)
  Interventions: Other: saline
- M-group (Experimental): patients receiving an IM Meloxicam injection near the nerve root (periradicular)
  Interventions: Drug: Meloxicam

INTERVENTIONS:
Other: saline — The patients received an IM injection of saline near the nerve root (periradicular)
  Arms: C-group
Drug: Meloxicam — The patients received an IM injection of meloxicam near the nerve root (periradicular)
  Other Names: mobic
  Arms: M-group

SUMMARY:
This randomized, double-blind, placebo control, cross-over study tested the hypothesis that periradicular injections of Meloxicam would reduce recent onset low back pain and improve physical activity compared to saline injection at 3 months follow-up evaluation

DETAILED DESCRIPTION:
In the present study we use a well-known non steroidal anti-inflammatory drug, meloxicam, in a novel way, an IM administration near a nerve root.

ELIGIBILITY:
Inclusion Criteria:

* low back pain from 6 months or less
* older than 18 years

Exclusion Criteria:

* not able to understand and sign the written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline NRS pain scale score at different consecutive follow up assessments | 5 minutes, 1, 6, 12 and 24 hours, 1, 5, 15, 30 and 90 days
  Patients reported a numeric value to evaluate pain (0= no pain, 10= wrost pain)

SECONDARY OUTCOMES:
Change from baseline level of physical activities and life quality at different consecutive follow up yes/no questionnaire | 5 minutes, 1, 6,12 and 24 hours, 1, 5, 15, 30 and 90 days
  pain-related insomnia, physical assistance, sport activities, work absence were assessed using a structured questionnaire with dichotomous items (yes/no presence of impairment to the selected item)

CONTACTS AND LOCATIONS:
Overall Officials: battista borghi, MD, Prof, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borghi B, Aurini L, White PF, Mordenti A, Lolli F, Borghi R, Martignani M, Greggi T. Long-lasting beneficial effects of periradicular injection of meloxicam for treating chronic low back pain and sciatica. Minerva Anestesiol. 2013 Apr;79(4):370-8. Epub 2013 Jan 10. PMID 23306395
- [Background] Aurini L, Borghi B, White PF, TOGNu A, Rossi B, Fini G, Fusco P, Mosca M, Borghi R. Treatment of chronic cervicobrachial pain with periradicular injection of meloxicam. Minerva Anestesiol. 2016 Apr;82(4):411-8. Epub 2015 Sep 3. PMID 26337371